CLINICAL TRIAL: NCT02930356
Title: Effects of Nonsurgical Periodontal Therapy on Plasma Hepatocyte Growth Factor Levels in Smokers and Non Smokers With Chronic Periodontitis
Brief Title: Effect of Tooth Cleaning in Smokers and Non Smokers With Gum Disease.
Acronym: ETCSNSGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, C.BHARGAVI, PG STUDENT, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D149206028
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSPT-Test group (Experimental): NSPT was done after administration of pre procedural mouth rinse in the test group (20 smokers with chronic periodontitis).Clinical parameters (GI,PI) were assessed at baseline and at the end of 3 months.2 ml blood was drawn to asses the plasma hepatocyte growth factor levels at baseline and at the end of 3 months.
  Interventions: Other: NSPT
- Scaling and root planing-Control group (Experimental): Scaling and root planing was done after administration of pre procedural mouth rinse in the control group (20 non smokers with chronic periodontitis).Clinical parameters (GI,PI) were assessed at baseline and at the end of 3 months.2 ml blood was drawn to asses the plasma hepatocyte growth factor levels at baseline and at the end of 3 months.
  Interventions: Other: Scaling and root planing

INTERVENTIONS:
Other: NSPT — NSPT was done by ultrasonic scalers after administration of pre procedural mouth rinse in the test group (20 smokers with chronic periodontitis).Clinical parameters (GI,PI) were assessed at baseline and at the end of 3 months.2 ml blood was drawn to assess the plasma hepatocyte growth factor levels at baseline and at the end of 3 months.
  Arms: NSPT-Test group
Other: Scaling and root planing — Scaling and root planing was done by ultrasonic scalers after administration of pre procedural mouth rinse in the control group (20 non smokers with chronic periodontitis).Clinical parameters (GI,PI) were assessed at baseline and at the end of 3 months.2 ml blood was drawn to assess the plasma hepatocyte growth factor levels at baseline and at the end of 3 months.
  Arms: Scaling and root planing-Control group

SUMMARY:
This study is intended to measure hepatocyte growth factor levels in smokers and non smokers with periodontitis before and after non surgical periodontal therapy.

DETAILED DESCRIPTION:
The study was randomised prospective,interventional clinical trial. The sample size for the study was 40 individuals aged between 20 to 60 years,equally divided into two groups.

Group l - smokers with chronic periodontitis (test) group. Group ll - non smokers with chronic periodontitis (controls)

At baseline both the groups were analysed for clinical and biochemical parameters and underwent non surgical periodontal therapy( scaling and root planning). All parameters were reassesed after 3 months.

A total of 40 patients( 20 somkers and 20 non smokers) from the outpatient wing of department of periodontics, Panineeya mahavidyalaya institute of dental sciences and research centre diagnosed with chronic periodontitis and willing to participate in the study.

Clicical parameters included gingival index and periodontal index. Biochmeical parameters included plasma hepatocyte growth factor.

ELIGIBILITY:
Inclusion Criteria:

* probing depth >4mm
* clinical attachment loss>2mm

Exclusion Criteria:

* patients younger than 20 years and greater than 60 years
* presence of any chronic conditions like diabetes,infections
* antibiotic therapy received preceeding 3 months
* former smokers who had quit the habit of smoking
* patients who already underwent periodontal therapy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome of the study was to measure plasma heaptocyte growth factor level | baseline, 3 months
  The change in plasma hepatocyte growth factor level was measured at baseline and at the end of 3 months after scaling and root planing.2 ml blood was drawn from the patient to assess the hepatocyte growth factor levels.biochemical analysis was done by ELISA test i.e., blood samples from both smokers and non smokers with chronic periodontitis were taken at baseline and at the end of 3 monthd

SECONDARY OUTCOMES:
gingival index | baseline and 3 months
  The secondary outcome of the study is to measure gingival index at baseline and 3 months after scaling and root planing. gingival index was assesed using williams periodontal probe
periodontal index | baseline and 3 months
  The secondary outcome of the study is to measure periodontal index at baseline and 3 months after scaling and root planing. periodontal index was assesed using williams periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Veerendranath R Panthula, MDS, Study Director — Panineeya Mahavidyalaya Institute of Dental Sciences and Research Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anil S, Vellappally S, Preethanath RS, Mokeem SA, AlMoharib HS, Patil S, Chalisserry EP, Al Kheraif AA. Hepatocyte growth factor levels in the saliva and gingival crevicular fluid in smokers with periodontitis. Dis Markers. 2014;2014:146974. doi: 10.1155/2014/146974. Epub 2014 Oct 15. PMID 25389376
- [Background] Rudrakshi C, Srinivas N, Mehta DS. A comparative evaluation of hepatocyte growth factor levels in gingival crevicular fluid and saliva and its correlation with clinical parameters in patients with and without chronic periodontitis: A clinico-biochemical study. J Indian Soc Periodontol. 2011 Apr;15(2):147-51. doi: 10.4103/0972-124X.84384. PMID 21976839